CLINICAL TRIAL: NCT04890925
Title: Evaluating The Effectiveness Of A Community Support Network Intervention For
Brief Title: A Community Support Network Intervention in SOAR Project Intimate Partner Violence-Related Traumatic Brain Injury
Acronym: SOAR-CSNI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: BrainTrust Canada (Unknown); The Kelowna Women's Shelter (Unknown); ABI Wellness (Unknown); Nanaimo Brain Injury Society (Unknown)
Responsible Party: Principal Investigator, Paul van Donkelaar, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H20-02412
Record Dates: First submitted 2021-05-05; First posted 2021-05-18 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Brain injury; Cognitive functions; Domestic violence; Intimate partner violence; Quality of life; Strangulation; Women
MeSH Terms: conditions — Brain Concussion; Brain Injuries | interventions — Methods

STUDY DESIGN:
Intervention Model Description: This is an experimental design. A comparison with control group is made to evaluate time related changes. The intervention (Community Support Network) group will be compared with a group receiving usual care to investigate 6 months intervention-induced effect.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Women who have experienced intimate partner violence but no sustained brain injury (Brain Injury Severity Assessment; BISA = 0)
- Community Support Network (CSN) intervention group (Experimental): The SOAR Community Support Network (CSN) intervention includes cognitive training, aerobic exercise, mindfulness meditation, counselling, quality of life tracking.
  Interventions: Behavioral: Community Support Network (CSN) intervention
- Usual care (Active Comparator): Participants in this group will receive dose-equivalent usual care
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Community Support Network (CSN) intervention — The SOAR Community Support Network (CSN) intervention is a multi-pillar, interdisciplinary system platform focused on improving higher order cognitive functions through aerobic exercise, mindfulness meditation, counselling, quality of life tracking, and cognitive exercises. The goal is to improve cognitive functions such as executive function, reasoning, and memory among those experiencing the effects of brain injury. Individually tailored protocol is administered to each participant. Goals are set daily, weekly, and monthly, and accomplishments tracked in a database. The CSN seeks to test and evaluate the success of the program when applied, and tailored, to survivors of brain injury in intimate partner violence.
  Other Names: Behavioral training; Cognitive and physical training
  Arms: Community Support Network (CSN) intervention group
Behavioral: Usual care — Participants in this group will receive dose-equivalent usual care based on the findings of a recent survey of the Canadian Rehabilitation Clinicians for concussion management, scoping review and clinical studies. Based on the evidence, usual care in this study will consist of education and aerobic exercises. Education includes information about the injury, recovery, management, nutrition, hydration, sleep, reassurance and goal setting that will be adapted to make appropriate to the population of this study. Aerobics include stationary cycling and treadmill exercises.
  Arms: Usual care

SUMMARY:
Intimate Partner Violence (IPV) comprises physical, sexual and emotional abuse and controlling behaviors imposed by an intimate partner. It is estimated that up to 92% of women who survive IPV may have suffered one or more traumatic brain injuries (TBI) from blows to the head, face, and neck, and/or anoxia or hypoxia due to strangulation. Even mild TBI may manifest as alternations in consciousness, black out, dizziness, disorientation, anxiety, depression, post-traumatic stress disorder, muscles weakness or paralysis and deficits in memory, attention, planning as well as executive functions. These signs and symptoms of TBI and their consequences impact the quality of life of women surviving IPV. Furthermore, survivors experiencing multiple IPV may acquire larger extent of the injury. Though this is recognized as an urgent and serious issue worldwide, it has been remarkably understudied.

To improve the quality of life of women experiencing IPV-related TBI, and to prevent potential longer-term consequences, an evidence-based therapeutic treatment is an urgent need. The Supporting Survivors of Abuse and Brain Injury through Research (SOAR) Project at the University of British Columbia-Okanagan was designed to integrate TBI knowledge into community-based supports. This Michael Smith Foundation for Health Research (MSFHR) trainee application will focus on the evaluation of the effectiveness of a community support network intervention for women with IPV-related TBI. The outcomes will generate valuable evidence to inform potential new TBI-informed policies regarding community-based and health care supports for survivors of IPV.

DETAILED DESCRIPTION:
Globally, about 35% of women experience intimate partner violence (IPV) over the course of their lives. The COVID-19 pandemic has resulted in a rapid increase of the incidence of IPV as vulnerable women are more likely to be trapped at home with their abusers. In Canada, IPV affects one in four women over their lifetime. In a study conducted in the United States, a heterogeneous (with respect to race, age, education level and employment status) sample of 99 community and shelter women, showed that about 75% sustained at least one IPV-related traumatic brain injury (TBI) and 50% of women sustained multiple IPV-related TBIs. Similar to post-concussive signs and symptoms, women with IPV-related TBI demonstrate cognitive impairments (e.g., deficits in memory, attention, reasoning, planning and executive functioning), psychopathological problems (such as depression, anxiety, fatigue and post-traumatic stress disorders), and/or sensorimotor problems (such as paralysis or paresis of facial or extremity muscles, numbness, loss of sensation, muscle spasms, facial droop, and unilateral weakness), due to blows to the head, face, or neck and/or strangulation which ultimately impacts quality of life.

The very few studies conducted in this population have reported the prevalence of IPV-related TBI, characteristic signs and symptoms, prevalence and primary sequelae of non-fatal strangulation, and brain network organization associated with TBI and its cognitive effects. A recent randomized trial on prevention of IPV and relationship problems focused on the parents of newborns demonstrated that prevention interventions for at-risk couples were not effective and rather showed iatrogenic effects for some couples. Therefore, therapeutic treatment for IPV-related TBI survivors is crucial, and any physical or cognitive impairment in these survivors require therapeutic interventions similar to non-partner related TBIs.

Effective therapeutic interventions would not only improve IPV-related TBI survivors' quality of life but also has the potential to prevent longer-term neurodegeneration if early detection is possible and timely treatment is provided. However, women rarely receive any therapeutic assessment or interventions after sustaining IPV-related TBI due to the lack of awareness regarding early detection and need of therapeutic interventions. On the other hand, evidence-based therapeutic interventions to improve the quality of life of survivors of IPV-related TBI are still lacking.

The Supporting Survivors of Abuse and Brain Injury through Research (SOAR) Project at UBC-Okanagan is a multidisciplinary, community-based partnership designed to i) investigate the incidence and characteristics of IPV-related TBI; ii) use integrated knowledge translation to co-create and disseminate knowledge products designed to increase knowledge and awareness of TBI in those who provide support for IPV survivors; and iii) evaluate the effectiveness of a community support network intervention for women with IPV-related TBI. This MSFHR trainee application will focus on this last aim.

This project will characterize quality of life, resilience, and neurocognitive and sensorimotor function prior to, immediately after, and 6 months after a 6-month community-based intervention incorporating executive function, physical activity, mindfulness/meditation, and health counseling components by comparing with a group receiving usual care and control participants. In addition, exploratory analyses will demonstrate the response to the intervention depending upon the severity of the IPV-related TBI, whether strangulation was part of the experience or not, and the extent of psychopathological comorbidities (e.g., post traumatic stress disorders, anxiety, depression, adverse childhood experiences, etc.).

This study aims to disseminate the findings not only through conference presentations and peer-reviewed journal publications but also through ongoing engagement with our local, regional, and national community partner organizations. We have already co-developed and implemented a knowledge product - the Women's Support Workers module of the Concussion Awareness Training Tool (CATT) to help raise knowledge and awareness of brain injury in those who provide support to survivors of IPV. We would envision incorporating some of the key takeaway findings from the SOAR project into an updated version of the CATT module.

The expected outcomes of this study will add strong evidence to the effectiveness of therapeutic interventions for, and strengthen our understanding of, this understudied experience. More broadly, this study will (i) enhance professional knowledge and research skills in understanding this underserved population, (ii) build up research knowledge on this topic, and (iii) increase knowledge on the efficacy of a novel intervention. Thus, clearly and objectively characterizing the potential for a community support network to improve resiliency, quality of life, and neurocognition will have far-reaching implications for social support policy and funding for this population and their caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Participants who identify as women and are survivors of IPV-related TBI

Exclusion Criteria:

* Pregnancy; any diagnosed neurological disorder other than brain injury known to affect cerebrovascular, neurocognitive, and/or sensorimotor function (e.g., stroke, Parkinson's, Alzheimer's, cerebral palsy, multiple sclerosis, migraine, seizures, etc.); taking any medication that might alter your blood pressure; have an injury or illness which affects your joints like arthritis. Participants will be tested in the early follicular phase or, if on combined hormonal contraception, at the end of the week that is off this contraception.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Cambridge Brain Science tasks (Now called Creyos) for assessing change in neuroconginitve functions and Task Switching Task for assessing executive functions | The 1st and 2nd sessions (one month apart) will occur prior to the enrollment to the intervention, the 3rd within 3 days of completing the intervention, and the 4th, 6 months after completing the intervention.
  Two purposes.
  1. To measure "change" from baseline at one month.
  2. To measure intervention-induced change, immediately after intervention and at 6 months post intervention
  Assessments include 12 different tasks to measure short-term memory, response inhibition, attention, verbal reasoning, visuospatial working memory, deductive reasoning, episodic memory, visuospatial processing, mental rotation, planning, spatial short-term memory, and working memory. The detail on CBS tests are available online at https://cambridgebrainsciences.com. Some of the tasks have to be solved as quickly and accurately as possible, whereas others have to be solved only as accurately as possible. Neurocognitive functions are assessed in terms of accuracy (number of correct judgments) and efficiency (ratio between total judgments and correct judgments) and/or speed (number of judgments at all) for each subtest. Higher scores indicate higher performance in each task.
Connor-Davidson Resiliency Scale to measure change in resilience | The 1st and 2nd sessions (one month apart) will occur prior to the enrollment to the intervention, the 3rd within 3 days of completing the intervention, and the 4th, 6 months after completing the intervention.
  Two purposes.
  1. To measure "change" from baseline at one month.
  2. To measure intervention-induced change, immediately after intervention and at 6 months post intervention
  Resiliency will be characterized using the Connor-Davidson Resilience Scale. This 25-item self-rated questionnaire measures responses to five factors associated with resilience on a 5-point Likert scale as follows: not true at all (0), rarely true (1), sometimes true (2), often true (3), and true nearly all of the time (4). The scale is rated based on how the participant has felt over the past month. The total score ranges from 0-100, with higher scores reflecting greater resilience. It has sound psychometric properties.

SECONDARY OUTCOMES:
Medical Outcomes study Questionnaire Short Form 36 (SF-36) to measure change in overall health status. | The 1st and 2nd sessions (one month apart) will occur prior to the enrollment to the intervention, the 3rd within 3 days of completing the intervention, and the 4th, 6 months after completing the intervention.
  Two purposes.
  1. To measure "change" from baseline at one month.
  2. To measure intervention-induced change, immediately after intervention and at 6 months post intervention
  Quality of Life will be measured using a modified version of the SF-36. This 36-item questionnaire consists of 8-scaled scores covering several aspects of quality of life and general health. The SF-36 has eight scaled (Vitality, Physical functioning, Bodily pain, General health perceptions, Physical role functioning, Emotional role functioning, Social role functioning, and Mental health) scores. The scores are weighted sums of the questions in each section. Scores range from 0 - 100; with lower scores indicating more disability and higher scores indicating less disability. The SF-36 is a reliable and well validated tool.

CONTACTS AND LOCATIONS:
Overall Officials: Kelsey Helm, Study Director — SOAR project at UBC
Locations (1):
- Nanaimo Brain Injury Society, Nanaimo, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided
There is a plan to make individual participant data available to other researchers. However, it has not been finalized.

REFERENCES:
- [Result] Buttell F, Ferreira RJ. The hidden disaster of COVID-19: Intimate partner violence. Psychol Trauma. 2020 Aug;12(S1):S197-S198. doi: 10.1037/tra0000646. Epub 2020 Jun 22. PMID 32567875
- [Result] Colantonio A. Beyond Football: Intimate Partner Violence and Concussion/Brain Injury. Canadian Psychology. 2020.
- [Result] Valera EM, Berenbaum H. Brain injury in battered women. J Consult Clin Psychol. 2003 Aug;71(4):797-804. doi: 10.1037/0022-006x.71.4.797. PMID 12924684
- [Result] Valera EM, Cao A, Pasternak O, Shenton ME, Kubicki M, Makris N, Adra N. White Matter Correlates of Mild Traumatic Brain Injuries in Women Subjected to Intimate-Partner Violence: A Preliminary Study. J Neurotrauma. 2019 Mar 1;36(5):661-668. doi: 10.1089/neu.2018.5734. Epub 2018 Oct 4. PMID 29873292
- [Result] Patch M, Anderson JC, Campbell JC. Injuries of Women Surviving Intimate Partner Strangulation and Subsequent Emergency Health Care Seeking: An Integrative Evidence Review. J Emerg Nurs. 2018 Jul;44(4):384-393. doi: 10.1016/j.jen.2017.12.001. Epub 2017 Dec 30. PMID 29292069
- [Result] Valera E, Kucyi A. Brain injury in women experiencing intimate partner-violence: neural mechanistic evidence of an "invisible" trauma. Brain Imaging Behav. 2017 Dec;11(6):1664-1677. doi: 10.1007/s11682-016-9643-1. PMID 27766587
- [Result] Smirl JD, Jones KE, Copeland P, Khatra O, Taylor EH, Van Donkelaar P. Characterizing symptoms of traumatic brain injury in survivors of intimate partner violence. Brain Inj. 2019;33(12):1529-1538. doi: 10.1080/02699052.2019.1658129. Epub 2019 Aug 23. PMID 31442093
- [Result] Heyman RE, Slep AMS, Lorber MF, Mitnick DM, Xu S, Baucom KJW, Halford WK, Niolon PH. A Randomized, Controlled Trial of the Impact of the Couple CARE for Parents of Newborns Program on the Prevention of Intimate Partner Violence and Relationship Problems. Prev Sci. 2019 Jul;20(5):620-631. doi: 10.1007/s11121-018-0961-y. PMID 30535623
- [Result] Kondo A, Shahpasand K, Mannix R, Qiu J, Moncaster J, Chen CH, Yao Y, Lin YM, Driver JA, Sun Y, Wei S, Luo ML, Albayram O, Huang P, Rotenberg A, Ryo A, Goldstein LE, Pascual-Leone A, McKee AC, Meehan W, Zhou XZ, Lu KP. Antibody against early driver of neurodegeneration cis P-tau blocks brain injury and tauopathy. Nature. 2015 Jul 23;523(7561):431-436. doi: 10.1038/nature14658. Epub 2015 Jul 15. PMID 26176913
- [Result] Iverson KM, Sayer NA, Meterko M, Stolzmann K, Suri P, Gormley K, Nealon Seibert M, Yan K, Pogoda TK. Intimate Partner Violence Among Female OEF/OIF/OND Veterans Who Were Evaluated for Traumatic Brain Injury in the Veterans Health Administration: A Preliminary Investigation. J Interpers Violence. 2020 Jul;35(13-14):2422-2445. doi: 10.1177/0886260517702491. Epub 2017 Apr 18. PMID 29294714
- [Result] Dobney DM, Miller MB, Tufts E. Non-pharmacological rehabilitation interventions for concussion in children: a scoping review. Disabil Rehabil. 2019 Mar;41(6):727-739. doi: 10.1080/09638288.2017.1400595. Epub 2017 Nov 20. PMID 29157025
- [Result] Varner CE. Specialized concussion clinic referrals are not intended for all acute concussion patients in the emergency department. CJEM. 2019 Nov;21(6):694-697. doi: 10.1017/cem.2019.430. No abstract available. PMID 31771689
- [Result] Varner CE, McLeod S, Nahiddi N, Lougheed RE, Dear TE, Borgundvaag B. Cognitive Rest and Graduated Return to Usual Activities Versus Usual Care for Mild Traumatic Brain Injury: A Randomized Controlled Trial of Emergency Department Discharge Instructions. Acad Emerg Med. 2017 Jan;24(1):75-82. doi: 10.1111/acem.13073. PMID 27792852
- [Result] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Result] Teel E, Brossard-Racine M, Corbin-Berrigan LA, Gagnon I. Perceptual Cognitive Training Does Not Improve Clinical Outcomes at 4 and 12 Weeks Following Concussion in Children and Adolescents: A Randomized Controlled Trial. J Head Trauma Rehabil. 2021 Mar-Apr 01;36(2):E97-E107. doi: 10.1097/HTR.0000000000000633. PMID 33201041